CLINICAL TRIAL: NCT02541344
Title: Double-blind, Randomised, Placebo-controlled, Three-way Crossover Clinical Investigation to Evaluate the Benefit of IQP-VV-102 in Reducing Postprandial Glucose Level in Overweight Caucasian Subjects
Brief Title: Benefit of IQP-VV-102 in Reducing Postprandial Glucose Level in Overweight Caucasian Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: INQ/024613
Record Dates: First submitted 2015-08-24; First posted 2015-09-04 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Prediabetes; Hyperglycemia
MeSH Terms: conditions — Prediabetic State; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose 1 of IQP-VV-102 (Active Comparator): Total 4 tablets (2 tablets with active ingredients and 2 placebo tablets) to be taken, 15 minutes before test meals (on 3 treatment days at the study site) with 200mL of water.
  Interventions: Device: Dose 1 of IQP-VV-102
- Dose 2 of IQP-VV-102 (Active Comparator): Total 4 tablets (4 tablets with active ingredients) to be taken, 15 minutes before test meals (on 3 treatment days at the study site) with 200mL of water.
  Interventions: Device: Dose 2 of IQP-VV-102
- Placebo (Placebo Comparator): Total 4 placebo tablets, 15 minutes before test meals (on 3 treatment days at the study site) with 200mL of water.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Dose 1 of IQP-VV-102 — Dose 1 (D1) group will take 2 tablets with active ingredients and 2 placebo tablets.
  Arms: Dose 1 of IQP-VV-102
Device: Dose 2 of IQP-VV-102 — Dose 2 (D2) group will take 4 tablets with active ingredients.
  Arms: Dose 2 of IQP-VV-102
Device: Placebo — Placebo group will take 4 placebo tablets.
  The placebo is designed to be identical to IQP-VV-102.
  Arms: Placebo

SUMMARY:
In this trial, the investigational product , the active ingredients which has been proven to reduce postprandial glucose in healthy and diabetic patients, will be tested. The primary aim of this clinical study is to evaluate the possibility of the investigational product to reduce the rise of postprandial glucose AUC level in overweight Caucasian subjects with normal to prediabetic biomarkers (IFG/HbA1C), without prompting a disproportionate rise in insulin levels.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* BMI between ≥ 25 and < 30 kg/m2
* Normal to prediabetic biomarkers: FBG 3.9-6.9 mmol/L / 70-125mg/dL and HbA1c 4-6.4%
* Willing to take test meal and adhere to consumptions of pre-prepared meals supplied (controlled by subject diary)
* Willing to maintain same level of physical activity during the study
* Willing to arrive at the study site with the same, non-strenuous means of transportation during the study
* Negative pregnancy testing (beta hCG) for women of childbearing potential during screening
* Women of child-bearing potential have to agree to use appropriate birth control methods during the study period
* Written informed consent of the subject to participate is a prerequisite for study participation

Exclusion Criteria:

* Known sensitivity to L-arabinose and grape marc extracts, or any sources of the active ingredients and excipients
* Use of medications or dietary supplements that may influence body weight 4 weeks, and gastrointestinal functions 2 weeks prior to enrolment and during the study
* Use of anti-diabetic medication
* Strenuous exercise within one day prior to blood glucose sampling (including screening).
* History of bariatric surgery, small bowel resection, or extensive bowel resection
* Difficult veins
* Recent blood donation in the last 1 month prior to study
* Pregnancy or nursing
* Clinically relevant excursions of safety parameters
* Any other serious condition or disease that renders subjects ineligible
* Smoking
* Exceeding safe alcohol consumption (men: ≥ 21 units/week; women: ≥ 14 units/week) and any alcohol consumption within 24 hours before venous blood glucose sampling
* All vegetarians and subjects with self-reported diet high in fat or protein
* Subjects are not able to communicate with local study staff
* Recent antibiotic and cortisone use up to one week and during the study
* Participation in another study during the last 30 days of the screening visit (V1)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Percentage change in raised postprandial glucose (PPG) AUC levels of the verum groups (dose D1 and dose D2) compared against the placebo among normal to prediabetic overweight Caucasian subjects. | 120 minutes
  Measures raised PPG AUC levels (mmol/L) from 0-120 minutes on each visit

SECONDARY OUTCOMES:
Change in incremental PPG AUC level (mmol/L) | 120 minutes
  Measured from 0-120 minutes after intake of verum or placebo on recruited subjects on each of the 3 visit days.
Change in total and incremental PPG AUC level (mmol/L) | 180 minutes
  Measured from 0th minute, to 60th, 90th and 180th minute after intake of verum or placebo on subjects on each of the 3 visit days.
Changes in PPG concentration | 180 minutes
  Measured at 15, 30, 45, 60, 90, and 120 minutes after intake of verum or placebo on recruited subjects on each of the 3 visit days.
Dose response of PPG level | Measured after intake of verum or placebo on recruited subjects on each of the 3 visit days.
Change in total and incremental AUC insulin level (mmol/L) | 180 minutes
  Measured from 0th minute to 120th and 180th minutes after intake of verum or placebo on recruited subjects on each of the 3 visit days.
Dose response of insulin level | Measured after intake of verum or placebo on recruited subjects on each of the 3 visit days.
Change in total and incremental AUC triglyceride level | 180 minutes
  Measured from 0-180 minutes after intake of verum or placebo on recruited subjects on each of the 3 visit days.
Global evaluation of tolerability both by investigator and subjects | Throughout the study (8-14 days)
  Global scaled evaluation with "very good", "good", "moderate" and "poor"
Incidence of adverse events (Safety parameters evaluation) | Throughout the study period (8-14 days)
  Eg. Liver Function Test, Lipid parameters, Renal Function Tests.
Reported adverse events | Throughout the whole study period (8-14 days)
  For any adverse event, the term of the event, intensity, duration, seriousness, frequency, outcome and assessment of causality with the investigational product will be documented in the Case Report Form (CRF)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, PhD, Principal Investigator — Charite
Locations (1):
- analyze & realize GmbH, Berlin, State of Berlin, Germany